CLINICAL TRIAL: NCT03157492
Title: Enhanced Aural Rehabilitation for Cochlear Implant Users Via Telerehab Technology
Brief Title: Aural Rehabilitation for Cochlear Implant Users Via Telerehab Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gallaudet University (Other)
Collaborators: Columbia University (Other); The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Diane Brewer, Co-Principal Investigator Research Audiologist, Gallaudet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2508; 90RE5020 (Other Grant/Funding Number: NIDILRR)
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Hearing Loss; Deafness
Keywords: Adult; Post-lingual; Auditory training; Communication strategies; Speech tracking; Speech recognition; Quality of Life
MeSH Terms: conditions — Hearing Loss; Deafness

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either AR Treatment or Active (Cognitive Training) Control Group. Participants are not told they are in the control group. After the final assessment (two-month post-treatment), control group participants are offered the AR treatment.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aural Rehabilitation Group (Experimental): The AR Group will receive six 90-minute sessions including auditory training, informational counseling, and communication strategies.
  Interventions: Behavioral: Aural Rehabilitation Group
- Cognitive Training Group (Sham Comparator): The Cognitive Training Group will receive six 90-minute sessions including training exercises (Ken-Ken, Sudoku, Crosswords, Word Search, Spot the Difference) to improve speed and accuracy.
  Interventions: Behavioral: Cognitive Training Group

INTERVENTIONS:
Behavioral: Aural Rehabilitation Group — Participants will complete sessions in their home or office via the internet. Sessions will include listening activities, informational counseling and communication strategies training. Three assessment appointments are required. The goal is to evaluate the benefit of training on performance with a cochlear implant.
  Arms: Aural Rehabilitation Group
Behavioral: Cognitive Training Group — The Cognitive Training Group will receive six 90-minute sessions including training exercises (Ken-Ken, Sudoku, Crosswords, Word Search, Spot the Difference) to improve speed and accuracy. Three assessment sessions are also required.
  Arms: Cognitive Training Group

SUMMARY:
This study evaluates the benefits of short-term training via telehealth for post-lingually deafened adult cochlear implant users. Half the participants will receive aural rehabilitation and the other half cognitive training. The hypothesis is that short-term aural rehabilitation via telerehab technology will improve outcomes for post-lingually deafened cochlear implant users

DETAILED DESCRIPTION:
Aural rehabilitation training (AR) has been demonstrated to improve outcomes for adult cochlear implant users. There are both financial and non-financial barriers to AR service delivery including accessibility (mobility, distance and transportation problems), accommodation (time off work impossible, caring for family) and availability (limited providers in rural areas, financial constraints, and lack of transportation. In this study the investigators will measure the impact of telerehab delivery on optimizing speech recognition, communication function, goals, social participation and hearing handicap.

Twenty-four participants will be randomly assigned to one of two treatment groups: aural rehabilitation (AR) and cognitive training (CT). Participants will complete six 90-minute treatment sessions in their home or office via a telerehab platform. Participants will come to a center for three 90-minute assessment sessions: pre-treatment, 1 week, and 2 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Speech Tracking rate of at least 20 words per minute
* Sentence recognition scores (CasperSent) between 10% and 85%
* Passing score on cognitive screener (Callahan et al., 2002)

Exclusion Criteria:

* Less than 18 years of age
* Pre-lingually deafened
* Prior Aural Rehabilitation with cochlear implant
* Greater than three years post-activation of CI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2021-10-13 (Actual)

PRIMARY OUTCOMES:
Change in Sentence Recognition CasperSent (Boothroyd, 2008) | Pre-training, One-week and Two-months post-training
  Percent correct scores on CasperSent topic-related recorded sentences.

SECONDARY OUTCOMES:
Change in Client Oriented Scale of Improvement (COSI) (Dillon, James & Ginis, 1997) | Pre-training, One-week and Two-months post-training
  Participant rates hearing ability and degree of change due to treatment for three self- selected listening situations most important to them.
Change in Hearing Handicap Inventory (HHI) (Ventry & Weinstein,1982) | Pre-training, One-week and Two-months post-training
  Participant rates 25 statements as true Always, Sometimes, or Never. Two subscales are Emotional and Social/situational.
Change in Glasgow Benefit Inventory (GBI) (Robinson et al.,1996 | One-week and Two-months post-training
  Participant rates change statements of change post-treatment.
Change in Nijmegen Cochlear Implant Questionnaire (NCIQ) (Hinderdink et al., 2000) | Pre-training, One-week and Two-months post-training
  60-item questionnaire with three domains: Physical, Social and Psychological.

CONTACTS AND LOCATIONS:
Overall Officials: Diane M Brewer, MA, Principal Investigator — Gallaudet University; Claire M Bernstein, PhD, Principal Investigator — Gallaudet University
Locations (5):
- United States (5):
  - Gallaudet University, Washington D.C., District of Columbia
  - University of South Florida, Tampa, Florida
  - University of Maryland, College Park, Maryland
  - Columbia University, New York, New York
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boothroyd, A. CasperSent: A program for computer-assisted speech perception testing and training at the sentence level. J Am Acad Rehab Audiol. 2008;41:30-50.
- [Background] Callahan CM, Unverzagt FW, Hui SL, Perkins AJ, Hendrie HC. Six-item screener to identify cognitive impairment among potential subjects for clinical research. Med Care. 2002 Sep;40(9):771-81. doi: 10.1097/00005650-200209000-00007. PMID 12218768
- [Background] Dillon H, James A, Ginis J. Client Oriented Scale of Improvement (COSI) and its relationship to several other measures of benefit and satisfaction provided by hearing aids. J Am Acad Audiol. 1997 Feb;8(1):27-43. PMID 9046067
- [Background] Hinderink JB, Krabbe PF, Van Den Broek P. Development and application of a health-related quality-of-life instrument for adults with cochlear implants: the Nijmegen cochlear implant questionnaire. Otolaryngol Head Neck Surg. 2000 Dec;123(6):756-65. doi: 10.1067/mhn.2000.108203. PMID 11112975
- [Background] Robinson K, Gatehouse S, Browning GG. Measuring patient benefit from otorhinolaryngological surgery and therapy. Ann Otol Rhinol Laryngol. 1996 Jun;105(6):415-22. doi: 10.1177/000348949610500601. PMID 8638891
- [Background] Ventry IM, Weinstein BE. The hearing handicap inventory for the elderly: a new tool. Ear Hear. 1982 May-Jun;3(3):128-34. doi: 10.1097/00003446-198205000-00006. PMID 7095321